CLINICAL TRIAL: NCT03322202
Title: Training Therapists in Motivational Interviewing to Enhance Rehabilitation Participation for Spinal Cord Injury (SCI)
Brief Title: Training Therapists in Motivational Interviewing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Linda Ehrlich-Jones, Assistant Director of Center for Rehabilitation Outcomes Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 441247
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Motivational Interviewing
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group will be exposed to a Physical or Occupational Therapist trained in Motivational Interviewing. The control group will receive standard therapy communication.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient participants will be blinded as will an assessor measuring participation during sessions. Therapist participants will be aware of the arm in which they will be placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Physical and Occupational Therapists will have 16 hours of training in Motivational Interviewing and use these techniques during sessions with patients.
  Interventions: Behavioral: Motivational Interviewing
- Control (No Intervention): Therapists will not participate in additional training.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing is a communication style that is intended to give patients the tools to reach goals through their own desires and actions.
  Arms: Motivational Interviewing

SUMMARY:
The purpose of this study is to test the efficacy of a Motivational Interviewing intervention on therapy participation as performed by physical and occupational therapists in an inpatient setting with patients with spinal cord injuries.

DETAILED DESCRIPTION:
Physical and Occupational Therapists that work in the inpatient spinal cord injury unit will be trained in Motivational Interviewing and will use the communication style to determine whether it is an effective tool to increase participation in therapy as opposed to patients who will have Physical and Occupational Therapists that are not trained in Motivational Interviewing.

ELIGIBILITY:
Therapist Inclusion Criteria:

* Inpatient therapist specializing in spinal cord injury patients for at least 3 months
* Practicing on one of the two designated inpatient units
* Willing to collect Patient Rehabilitation Participation Scale (PRPS) daily on their patients
* Willing to audio record conversations with patients;
* Willing and able to participate in 16 hours of MI training
* Willing to receive feedback on MI skills

Therapist Exclusion Criteria:

* Inpatient therapist specializing in spinal cord injury patients for less than 3 months
* Unwilling or unable to follow the study protocol

Patient Inclusion Criteria:

* Inpatient in the spinal cord injury unit
* Has a physical or occupational therapist who is a participant in the study

Patient Exclusion Criteria:

* Unwilling to allow for therapy sessions to be recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Increased therapy participation | 4 weeks
  To measure therapy participation in inpatients with SCI treated by rehabilitation therapists trained in Motivational Interviewing (MI) compared to those treated by therapists not trained to use MI

SECONDARY OUTCOMES:
Treatment Satisfaction | 4 weeks
  To measure treatment satisfaction in inpatients with SCI treated by rehabilitation therapists trained in MI compared to those treated by therapists not trained to use MI
Self-care and mobility | 4 weeks
  To measure Inpatient Rehabilitation Facility (IRF)-Patient Assessment Instrument (PAI) efficiency in the domains of self-care and mobility in inpatients with SCI treated by rehabilitation therapists trained in MI compared to those treated by therapists not trained to use MI
Efficacy of Motivational Interviewing (MI) Training | 4 weeks
  To measure the efficacy of MI training by measuring adherence to MI counseling skills in rehabilitation therapists trained to use MI compared to those not trained to use MI

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ehrlich-Jones, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan Abilitylab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teeter L, Gassaway J, Taylor S, LaBarbera J, McDowell S, Backus D, Zanca JM, Natale A, Cabrera J, Smout RJ, Kreider SE, Whiteneck G. Relationship of physical therapy inpatient rehabilitation interventions and patient characteristics to outcomes following spinal cord injury: the SCIRehab project. J Spinal Cord Med. 2012 Nov;35(6):503-26. doi: 10.1179/2045772312Y.0000000058. PMID 23318034
- [Background] Lenze EJ, Munin MC, Quear T, Dew MA, Rogers JC, Begley AE, Reynolds CF 3rd. The Pittsburgh Rehabilitation Participation Scale: reliability and validity of a clinician-rated measure of participation in acute rehabilitation. Arch Phys Med Rehabil. 2004 Mar;85(3):380-4. doi: 10.1016/j.apmr.2003.06.001. PMID 15031821
- [Background] Maclean N, Pound P. A critical review of the concept of patient motivation in the literature on physical rehabilitation. Soc Sci Med. 2000 Feb;50(4):495-506. doi: 10.1016/s0277-9536(99)00334-2. PMID 10641802
- [Background] Lundahl B, Kunz C, Brownell C, Tollefson D, Burke B. A meta-analysis of motivational interviewing: Twenty-five years of empirical studies. Research on Social Work Practice. 2010;20(2):137-160.
- [Background] Soderlund LL, Madson MB, Rubak S, Nilsen P. A systematic review of motivational interviewing training for general health care practitioners. Patient Educ Couns. 2011 Jul;84(1):16-26. doi: 10.1016/j.pec.2010.06.025. Epub 2010 Jul 25. PMID 20667432
- [Background] Bombardier CH, Ehde DM, Gibbons LE, Wadhwani R, Sullivan MD, Rosenberg DE, Kraft GH. Telephone-based physical activity counseling for major depression in people with multiple sclerosis. J Consult Clin Psychol. 2013 Feb;81(1):89-99. doi: 10.1037/a0031242. PMID 23379265
- [Background] Bombardier CH, Rimmele CT. Alcohol use and readiness to change after spinal cord injury. Arch Phys Med Rehabil. 1998 Sep;79(9):1110-5. doi: 10.1016/s0003-9993(98)90180-0. PMID 9749693
- [Background] Watkins CL, Auton MF, Deans CF, Dickinson HA, Jack CI, Lightbody CE, Sutton CJ, van den Broek MD, Leathley MJ. Motivational interviewing early after acute stroke: a randomized, controlled trial. Stroke. 2007 Mar;38(3):1004-9. doi: 10.1161/01.STR.0000258114.28006.d7. Epub 2007 Feb 15. PMID 17303766
- [Background] Ehrlich-Jones L, Mallinson T, Fischer H, Bateman J, Semanik PA, Spring B, Ruderman E, Chang RW. Increasing physical activity in patients with arthritis: a tailored health promotion program. Chronic Illn. 2010 Dec;6(4):272-81. doi: 10.1177/1742395309351243. Epub 2010 Aug 9. PMID 20696695
- [Background] O'Halloran PD, Blackstock F, Shields N, Holland A, Iles R, Kingsley M, Bernhardt J, Lannin N, Morris ME, Taylor NF. Motivational interviewing to increase physical activity in people with chronic health conditions: a systematic review and meta-analysis. Clin Rehabil. 2014 Dec;28(12):1159-71. doi: 10.1177/0269215514536210. Epub 2014 Jun 18. PMID 24942478
- [Background] Vong SK, Cheing GL, Chan F, So EM, Chan CC. Motivational enhancement therapy in addition to physical therapy improves motivational factors and treatment outcomes in people with low back pain: a randomized controlled trial. Arch Phys Med Rehabil. 2011 Feb;92(2):176-83. doi: 10.1016/j.apmr.2010.10.016. PMID 21272712
- [Background] Brodie DA, Inoue A, Shaw DG. Motivational interviewing to change quality of life for people with chronic heart failure: a randomised controlled trial. Int J Nurs Stud. 2008 Apr;45(4):489-500. doi: 10.1016/j.ijnurstu.2006.11.009. Epub 2007 Jan 26. PMID 17258218
- [Background] Tse MM, Vong SK, Tang SK. Motivational interviewing and exercise programme for community-dwelling older persons with chronic pain: a randomised controlled study. J Clin Nurs. 2013 Jul;22(13-14):1843-56. doi: 10.1111/j.1365-2702.2012.04317.x. Epub 2013 Jan 2. PMID 23279630
- [Background] Cowan RE, Nash MS, Anderson KD. Exercise participation barrier prevalence and association with exercise participation status in individuals with spinal cord injury. Spinal Cord. 2013 Jan;51(1):27-32. doi: 10.1038/sc.2012.53. Epub 2012 May 15. PMID 22584283
- [Background] Pellatt GC. Patient-professional partnership in spinal cord injury rehabilitation. Br J Nurs. 2004 Sep 9-22;13(16):948-53. doi: 10.12968/bjon.2004.13.16.15966. PMID 15389135
- [Background] Wiprovnick AE, Kuerbis AN, Morgenstern J. The effects of therapeutic bond within a brief intervention for alcohol moderation for problem drinkers. Psychol Addict Behav. 2015 Mar;29(1):129-35. doi: 10.1037/a0038489. Epub 2015 Feb 2. PMID 25642584
- [Background] Zuckoff A. "Why won't my patients do what's good for them?" Motivational interviewing and treatment adherence. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):514-21. doi: 10.1016/j.soard.2012.05.002. Epub 2012 May 4. PMID 22704048
- [Background] Pegg PO, Auerbach SM, Kiesler DJ, Plybon LE, Seel RT, Buenaver LF. The Impact of Patient-Centered Information on Patients' Treatment Satisfaction and Outcomes in Traumatic Brain Injury Rehabilitation. Rehabilitation Psychology. 2005;50(4):366-374.
- [Background] Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. Clin Psychol Psychother. 2010 May-Jun;17(3):231-9. doi: 10.1002/cpp.658. PMID 20013760
- [Background] Moyers TB, Martin T, Manuel JK, Hendrickson SM, Miller WR. Assessing competence in the use of motivational interviewing. J Subst Abuse Treat. 2005 Jan;28(1):19-26. doi: 10.1016/j.jsat.2004.11.001. PMID 15723728
- [Background] Miller WR, Rollnick S. Meeting in the middle: motivational interviewing and self-determination theory. Int J Behav Nutr Phys Act. 2012 Mar 2;9:25. doi: 10.1186/1479-5868-9-25. No abstract available. PMID 22385872
- [Background] Velasquez M, Maurer G, Crouch C, DiClemente C. Group treatment for substance abuse: A stages of change therapy book. New York: Guilford Press; 2001.
- [Background] Mead N, Bower P. Patient-centredness: a conceptual framework and review of the empirical literature. Soc Sci Med. 2000 Oct;51(7):1087-110. doi: 10.1016/s0277-9536(00)00098-8. PMID 11005395
- [Background] Lindberg J, Kreuter M, Person LO, Taft C. Patient Participation in Rehabilitation Questionnaire (PPRQ)-development and psychometric evaluation. Spinal Cord. 2013 Nov;51(11):838-42. doi: 10.1038/sc.2013.98. Epub 2013 Sep 17. PMID 24042990
- [Background] Lenze EJ, Munin MC, Quear T, Dew MA, Rogers JC, Begley AE, Reynolds CF. Significance of poor patient participation in physical and occupational therapy for functional outcome and length of stay. Arch Phys Med Rehabil. 2004 Oct;85(10):1599-601. doi: 10.1016/j.apmr.2004.03.027. PMID 15468017
- [Background] Miller WR, Yahne CE, Moyers TB, Martinez J, Pirritano M. A randomized trial of methods to help clinicians learn motivational interviewing. J Consult Clin Psychol. 2004 Dec;72(6):1050-62. doi: 10.1037/0022-006X.72.6.1050. PMID 15612851
- [Background] Hall AM, Ferreira PH, Maher CG, Latimer J, Ferreira ML. The influence of the therapist-patient relationship on treatment outcome in physical rehabilitation: a systematic review. Phys Ther. 2010 Aug;90(8):1099-110. doi: 10.2522/ptj.20090245. Epub 2010 Jun 24. PMID 20576715
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Mohr DC, Spring B, Freedland KE, Beckner V, Arean P, Hollon SD, Ockene J, Kaplan R. The selection and design of control conditions for randomized controlled trials of psychological interventions. Psychother Psychosom. 2009;78(5):275-84. doi: 10.1159/000228248. Epub 2009 Jul 11. PMID 19602916